CLINICAL TRIAL: NCT02387931
Title: SAGE: Supplementation in Adolescent Girls With Endometriosis
Brief Title: Supplementation in Adolescent Girls With Endometriosis
Acronym: SAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Stacey Missmer, Stacey Missmer, ScD, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P00007860
Record Dates: First submitted 2013-05-29; First posted 2015-03-13 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Endometriosis
Keywords: Adolescent; Endometriosis; Diet; Nutrition; Pain
MeSH Terms: conditions — Endometriosis; Pain | interventions — Cholecalciferol; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin D (Experimental): Vitamin D3 2000 IU daily taken for 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Fish Oil (Experimental): Fish Oil 1000 mg daily for 6 months
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): Placebo taken daily for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Nature Made Vitamin D 2000IU, 1 softgel taken daily
  Other Names: Nature Made Vitamin D 2000IU Liquid softgels
  Arms: Vitamin D
Dietary Supplement: Fish Oil — Nature Made ultra omega-3 mini fish oil 500mg, 2 soft gels taken daily
  Other Names: Nature Made ultra omega-3 mini fish oil 500mg, 2 daily
  Arms: Fish Oil
Other: Placebo — Placebo capsule, 2 taken daily
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether dietary supplementation with Vitamin D or Fish Oil can help to reduce physical and emotional symptoms in adolescent girls with endometriosis.

DETAILED DESCRIPTION:
This is a randomized controlled trial designed to evaluate the effect of dietary supplementation on endometriosis symptom remediation. Adolescent and young adults females aged 12 to 25 years with a surgically-confirmed diagnosis of endometriosis will be eligible for study participation. Subjects will be excluded if they have concurrent chronic illnesses that affect gastrointestinal absorption of nutrients (e.g., celiac disease, IBD, cystic fibrosis), a history of renal stones, are pregnant, or non-English speaking. Once consented, subjects will be randomized to one of 3 treatment assignments: 1) vitamin D3 2000 IU daily (n=30), 2) fish oil 1000 mg daily (n=30), 3) placebo (n=30) and will take these daily for 6 months. Baseline nutrient intake from food and supplements will be assessed using the Food Frequency Questionnaire (FFQ). The 142 item survey assesses usual dietary intake during the past year. Validated rating scales including the visual analog scale (VAS), SF-36, and the World Endometriosis EPHect questionnaires will be used to measure pain and overall quality of life. The SF-36 measures 8 health concepts relevant across disease groups, including limitations to physical or social activities because of health problems, vitality, and general health perception. Patients will complete a full review of medication usage, past medical history, family history, and other lifestyle factors. Anthropometrics will be measured, and vital signs obtained. Measures will be repeated at 3-month intervals for a total of 6 months. Blood will be drawn at baseline, and at 6 months to measure levels of fatty acids, vitamin D, parathyroid hormone (PTH), and calcium.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 12 years -25 years
* Previously surgically diagnosed at Boston Children's Hospital with endometriosis
* At least 6 weeks following laparoscopy
* Minimum pain score within the 4 weeks preceding study baseline
* Must be able to swallow an empty 00 gelatin capsule at baseline
* Must be willing to stop all vitamins and nutritional supplements during trial

Exclusion Criteria:

* Concurrent chronic illnesses that affect gastrointestinal absorption of nutrients (e.g., celiac disease, IBD, cystic fibrosis)
* Vitamin D level of greater than or equal to 100 ng/ml at study baseline
* History of renal stones
* No access to text messages or email
* Pregnancy
* Non-English speaking

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Endometriosis pain | 6 months
  Measured by change in the score of the visual analog scale (VAS) from baseline to 6 months.

SECONDARY OUTCOMES:
Quality of life | 6 months
  Measured by change in SF-36 and EPHect questionnaires from baseline to 6 months.
Pain medication usage | 6 months
  Measured via questionnaire of medication usage from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey A Missmer, ScD, Principal Investigator — Department of Reproductive Medicine, Brigham and Women's Hospital and Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nodler JL, DiVasta AD, Vitonis AF, Karevicius S, Malsch M, Sarda V, Fadayomi A, Harris HR, Missmer SA. Supplementation with vitamin D or omega-3 fatty acids in adolescent girls and young women with endometriosis (SAGE): a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2020 Jul 1;112(1):229-236. doi: 10.1093/ajcn/nqaa096. PMID 32453393